CLINICAL TRIAL: NCT04048954
Title: Prospective Study Evaluating the Impact of the Use of a Smartphone Application on the Detection of Complications Related to Smoking
Brief Title: Use of a Smartphone Application on the Detection of Complications Related to Smoking
Acronym: APPLITABAC
Status: Completed | Type: Observational
Sponsor: Weprom (Other)
Collaborators: Le Mans Town Hall (72) (Unknown); Department of Sarthe (72) (Unknown)
Responsible Party: Sponsor
Other Study IDs: WP-2019-01; NR1512030619 (Other: INDS)
Record Dates: First submitted 2019-07-30; First posted 2019-08-07 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2019-08

CONDITIONS: Tabagism; Lung Cancer; Chronic Obstructive Pulmonary Disease
Keywords: Screening; Tabagism; Chronic Obstructive Pulmonary Disease; Cancer; Lung
MeSH Terms: conditions — Lung Neoplasms; Pulmonary Disease, Chronic Obstructive; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- APPLITABAC arm: Use of a smartphone application on screening for complications related to tabagism
  Interventions: Device: Applitabac

INTERVENTIONS:
Device: Applitabac — Smartphone application in screening on tabagism complications

SUMMARY:
Smokers do not know the symptoms of cancer and wait on average 5 months with symptoms before consulting. 80% of lung cancers are diagnosed at too late and incurable stage.

Systematic CT screening of smokers is under evaluation and currently not supported because expensive and little used in real life (in the US 1.8% of smokers after 7 years of establishment in the USA).

An English study showed an increase in the number of operable stage cancers of 3% among smokers by calling them on a trailing cough by a simple poster campaign ("You smoke, you cough for more than 3 weeks, consult").

Regarding COPD, it is linked to tobacco in 85% of cases, affects 3.5 million French and is in 2013 the 4th leading cause of death in France. The evolution of COPD is marked by exacerbations, period of acute aggravation of symptoms, responsible for the deterioration of the quality of life or even hospitalization or death. COPD remains a silent killer responsible, according to this same summary review, of 16,500 deaths per year in France.

Dr DENIS has developed a web application that has shown a 7-month survival benefit by early detection of lung cancer relapses based on the reporting of patient symptoms analyzed by a validated algorithm in 300 patients and 1 randomized trial.

The Applitabac app takes this concept of symptom self-assessment by patients. By multiplying the number of symptoms analyzed compared to the English study, Applitabac should be able to increase the sensitivity of this early detection of COPD and increase the number of operable bronchial cancers and increase the chances of survival of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old
* Applitabac user who has received a notification directing him to his doctor
* Smoker or former smoker (current smoking cessation or ≤ 5 years)
* Patient informed of the use of his data and not opposing it

Exclusion Criteria:

* Presence of another evolutionary neoplasia in the past 2 years
* Patient who did not use the Applitabac app

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Smoker or former smoker
Sampling Method: Non-Probability Sample
Enrollment: 5671 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients fit for surgery for a symptomatic stage I-II lung cancer during the 12 weeks after the web-application rollout | 12 weeks
  Proportion of patients fit for surgery for a symptomatic stage I-II lung cancer during the 12 weeks after the web-application rollout

SECONDARY OUTCOMES:
Proportion of patients operated on for lung cancer during the first and second year of follow-up in comparaison of 2017/2018 | first and second year of follow-up
  Proportion of patients operated on for lung cancer during the first and second year of follow-up in comparaison of 2017/2018
Proportion of diagnosed lung cancers, by stage and total first and second year of follow-up | first and second year of follow-up
  Proportion of diagnosed lung cancers, by stage and total first and second year of follow-up
Stage of lung cancer surgery with Applitabac first and second year of follow-up | first and second year of follow-up
  Stage of lung cancer surgery with Applitabac first and second year of follow-up
Histological stage of diagnosed lung cancer | second year of follow-up
  Histological stage of diagnosed lung cancer
Stages of other cancers of Applitabac users diagnosed with Applitabac in the first and second year of follow-up | first and second year of follow-up
  Stages of other cancers of Applitabac users diagnosed with Applitabac in the first and second year of follow-up
Proportion of other cancers of Applitabac users diagnosed with Applitabac in the first and second year of follow-up | first and second year of follow-up
  Proportion of other cancers of Applitabac users diagnosed with Applitabac in the first and second year of follow-up
Proportion of Applitabac-induced thoracic interventions without a cancer diagnosis first and second year of follow-up | first and second year of follow-up
  Proportion of Applitabac-induced thoracic interventions without a cancer diagnosis first and second year of follow-up
Proportion of patients with another pathology detected by Applitabac in the first and second year of follow-up | first and second year of follow-up
  Proportion of patients with another pathology detected by Applitabac in the first and second year of follow-up
Stage of diagnosis of COPD detected by the application (GOLD classification : VEMS) | second year of follow-up
  Stage of diagnosis of COPD detected by the application (GOLD classification : VEMS)
Distribution of the stages of operated lung cancer, the two years preceding the implementation of Applitabac over similar periods | Two years before use of Applitabac
  Distribution of the stages of operated lung cancer, the two years preceding the implementation of Applitabac over similar periods
Compare the distribution of the stages of operated patients (app vs. not app) | second year of follow-up
  Compare the distribution of the stages of operated patients (app vs. not app)
Comparison of the stage distribution of patients operated before / after implementation of the application (via Epithor data base) | second year of follow-up
  Comparison of the stage distribution of patients operated before / after implementation of the application (via Epithor data base)
Number of users who want to quit after first use | 30 minutes after application implementation
  Number of users who want to quit after first use

CONTACTS AND LOCATIONS:
Locations (1):
- All MD, Le Mans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Denis F, Basch E, Septans AL, Bennouna J, Urban T, Dueck AC, Letellier C. Two-Year Survival Comparing Web-Based Symptom Monitoring vs Routine Surveillance Following Treatment for Lung Cancer. JAMA. 2019 Jan 22;321(3):306-307. doi: 10.1001/jama.2018.18085. PMID 30667494
- [Result] Ironmonger L, Ohuma E, Ormiston-Smith N, Gildea C, Thomson CS, Peake MD. An evaluation of the impact of large-scale interventions to raise public awareness of a lung cancer symptom. Br J Cancer. 2015 Jan 6;112(1):207-16. doi: 10.1038/bjc.2014.596. Epub 2014 Dec 2. PMID 25461805
- [Derived] Stavaux E, Goupil F, Barreau G, Septans AL, Dautzenberg B, Foulet-Roge A, Padilla N, Urban T, Denis F. Use of a Smartphone Self-assessment App for a Tobacco-Induced Disease (COPD, Cardiovascular Diseases, Cancer) Screening Strategy and to Encourage Smoking Cessation: Observational Study. JMIR Public Health Surveill. 2022 Feb 23;8(2):e19877. doi: 10.2196/19877. PMID 35195530